CLINICAL TRIAL: NCT01082653
Title: Phase I, Single Center, Prospective, Non-randomized, Open Label, Safety/Efficacy Study of the Infusion of Autologous Bone Marrow-derived Stem Cells, in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Safety/Efficacy Study for the Treatment of Amyotrophic Lateral Sclerosis
Acronym: ALS
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended due to lack of funding.
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-ALS-I
Record Dates: First submitted 2010-03-01; First posted 2010-03-08 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2013-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety (Experimental): infusion of autologous bone marrow-derived stem cells
  Interventions: Biological: autologous bone marrow-derived stem cells

INTERVENTIONS:
Biological: autologous bone marrow-derived stem cells — All patients will receive a unique one-time intrathecal infusion of the cell product suspended in infusion medium.

SUMMARY:
A Phase I, single center, prospective, non-randomized, open label, safety/efficacy study of the infusion of autologous bone marrow-derived stem cells, in 6 patients with Amyotrophic Lateral Sclerosis according to established criteria (1), (2) with a moderate to severe diagnosis of ALS according to the World Federation of Neurology El Escorial criteria.

The primary purpose of this study is to evaluate safety of the infusion procedure, as assessed by absence of complications at the site of infusion or the appearance of new neurologic deficit not attributed to the natural progression of the disease.

Secondary outcomes will include a)neurological evidence of trends toward a slowing down of the decline of the forced vital capacity (FVC) (3) and of the functional rating scale (ALS-FRS) scores, as assessed at 3-month intervals, b)evidence of a decline of the maximum voluntary isometric contraction-arm (MVIC-arm) and MVIC-grip Z (4) scores and c)patient evaluation that the treatment was effective and consider the possibility of a new cell product stem cell infusion.

Subjects who fulfill inclusion/exclusion criteria and sign informed consent will undergo an aspiration of bone marrow from the iliac crest for preparation of the cellular product.

The day of infusion, the investigational product will be injected into the patient's intrathecal space.

After cell infusion patients will be followed at WK 2, MN 1, MN 2, MN 6 and a long-term followup at MN 12 in the clinic and/or office. Electromyographic (EMG) studies, Forced vital capacity (FVC), functional rating scale (FRS) and maximum voluntary isometric contraction-arm (MVIC-arm) and MVIC-grip Z scores will have been used to assess the status of the disease before (historical record acceptable if done within three months of Screening Visit) and during the 12-month study period after cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects > 18 years of age.
2. Good understanding of the protocol and willingness to consent.
3. Moderate to severe Diagnosis of ALS according to the World Federation of Neurology El Escorial criteria.
4. Vital capacity at least 50% predicted value for gender, height and age.
5. More than 6 and less than 36 months of evolution of the disease.
6. Hematocrit greater than 30 % prior to bone marrow aspiration.
7. Platelet count greater than 100 Thousand/uL at screening.
8. INR less than or equal to 1.5.

Exclusion Criteria:

1. Any concurrent illness, which affects the bone marrow.
2. Any concomitant medication that affects the bone marrow.
3. Previous stem cell therapy.
4. Any lymphoproliferative disease.
5. Riluzole with 4 weeks of study entry and at any time during the study.
6. Hemophiliacs or subjects with bleeding disorders.
7. Known hypersensitivity to fetal bovine serum
8. HIV infection.
9. Serum creatinine > 3.0 in subjects not on hemodialysis.
10. Skin infection at the infusion site or systemic infection
11. Current smoker.
12. Active drug or alcohol addiction
13. Pregnant, planning to become pregnant or not on accepted birth control method if subject is of child bearing potential.
14. Subjects that are breast feeding.
15. Any condition that the Principal Investigator considers would render the subject unfit for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Safety | one year
  Safety of the infusion procedure, as assessed by absence of complications at the site of infusion or the appearance of new neurologic deficit not attributed to the natural progression of the disease.

SECONDARY OUTCOMES:
Efficacy | one year
  Neurological evidence of trends toward a slowing down of the decline of the forced vital capacity and of the functional rating scale scores, as assessed at 3 month intervals.
  Evidence of a decline of the maximum voluntary isometric contraction-arm (MVIC-arm) and MVIC-grip Z scores.
  Patient evaluation that the treatment was effective.

CONTACTS AND LOCATIONS:
Locations (1):
- TCA Cellular Therapy, Covington, Louisiana, United States